CLINICAL TRIAL: NCT07326618
Title: The Use of Virtual Reality Application in Improving Psychosocial Dysfunction in Schizophrenia
Brief Title: Cinematic Virtual Reality Intervention for Improving Psychosocial Functioning in Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Emine Ilgın Hoşgelen, Dr, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5297-GOA-2021/24-12
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; virtual reality; psychosocial functioning; social cognition; neurocognition; sense of presence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: The experimental group received received a cinematic virtual reality-based psychosocial intervention during 12 weeks on a weekly basis. The intervention consisted of different cinematic VR sessions delivered weekly. Sessions were designed to address psychosocial functioning, social interaction, and daily functioning. Participants continued to have their usual medical treatment.
  The control group also consisted of individuals with schizophrenia. Participants in this group did not receive the virtual reality intervention and they continued to receive treatment as usual throughout the study period.
  They participated in weekly face-to-face, non-interventional interviews during 12 weeks.
Masking Description: The rater of Personal and Social Performance Scale was blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinematic Virtual Reality Psychososcial Treatment Program Group (Experimental): Participants received cinematic VR sessions in this group on a weekly basis during 12 weeks
  Interventions: Behavioral: Cinematic Virtual Reality Psychososcial Treatment Program Group
- Control Group - Face to Face Interviews (No Intervention): This group consists of individuals with schizophrenia. Participants in this group did not receive the virtual reality intervention. They participated in weekly face-to-face, non-interventional interviews as part of treatment as usual for 12 weeks on a weekly basis.

INTERVENTIONS:
Behavioral: Cinematic Virtual Reality Psychososcial Treatment Program Group — cVR-PTP
  1. Week - Orientation to the Virtual Environment: Ability to use the VR headset, visual-spatial awareness related to the virtual environment
  2. Week - Orientation to the Virtual Environment: Ability to use the VR headset, visual-spatial awareness related to the virtual environment
  3. Week - Self-Care: Waking up in the morning, taking a shower
  4. Week - Social Interaction: Waiting at a crowded public transport stop, interacting with others
  5. Week - Mobility: Traveling with others on a tram
  6. Week - Mobility: Traveling with others on a ferry
  7. Week - Mobility and Daily Living Activities: Shopping at a traditional bazaar
  8. Week - Social Interaction: Going alone to a café
  9. Week - Daily Living Activities: Experiencing a grocery shopping
  10. Week - Independent Time Activities - Social Interaction: Participating in a cooking workshop
  11. Week - Social Interaction: watching aTV show with others
  12. Week - Social Interaction: Being in a pleasant family and friends setting
  Other Names: cVR-PTP
  Arms: Cinematic Virtual Reality Psychososcial Treatment Program Group

SUMMARY:
Virtual reality (VR) is a novel and innovative intervention method increasingly used in psychiatric research and treatment. VR allows individuals to experience realistic, everyday social situations in a safe and controlled environment. This study aims to examine the effects of a cinematic VR-based psychosocial intervention on individuals with schizophrenia who experience reduced psychosocial functioning and social isolation.

In this study, a Cinematic Virtual Reality Treatment Program (cVR-PTP) consisting of 12 weekly sessions was developed. Each session focuses on real-life social situations designed to support social interaction and daily functioning. The intervention aims to contribute to improvements in psychosocial functioning, social engagement, and overall functioning in individuals with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental disorder associated with significant impairments in psychosocial functioning. These impairments affect individuals' abilities to perform in daily life activities, maintain occupational functioning, and participate actively in social communities. Reduced psychosocial functioning is a major contributor to long-term disability in schizophrenia and is widely accepted as a core indicator of recovery beyond symptom remission.

Although antipsychotic medications are effective to a certain point in reducing positive symptoms, there is currently no pharmacological treatment that directly targets improvements in psychosocial functioning. For this reason, psychosocial interventions such as social skills training and social cognitive remediation programs have been developed to enhance social participation and functional outcomes in individuals with schizophrenia. However, these approaches often show limited effectiveness, and their benefits may not generalize to real-life situations or be equally effective for all patients.

Virtual reality (VR) has emerged as a promising alternative approach for psychosocial interventions in schizophrenia after the advances in technology. VR-based interventions allow individuals to engage in simulated social environments that offer ecological validity while maintaining a safe and controlled setting under the supervision of a mental health professional. Existing VR studies in schizophrenia have primarily based on computer-generated virtual environments or avatar-based characters.

In the present study, a cinematic virtual reality intervention program was created using 360-degree real world video recordings. This environmental seeting was designed to enhance immersion by presenting social situations as they naturally occur in everyday life. The study aimed to examine whether exposure to these cinematic VR scenarios could lead to improvements in psychosocial functioning in individuals with schizophrenia, compared to standard follow-up.

The objective of this study is to measure the effectiveness of cinematic basd VR for improving psychosocial functioning in schizophrenia by focusing on real-life-based immersive experiences. The other objective of this study is to measure the sense of presence of the partcipants in the cinematic virtual environment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stability over the past 12 weeks
* No changes in antipsychotic medication during last 6 monhts
* Having a score ≤70 on the PSP and and ≤61 on the Social and Occupational Functioning Assessment Scale (SOFAS)

Exclusion Criteria:

* Experienced a psychotic episode or suicide attempt in the past 12 weeks
* Received electroconvulsive therapy in the past 6 months
* Having a diagnosis of a serious physical or neurological disorder that could impact clinical functioning or sensory systems (visual or auditory), alcohol or substance use disorder, intellectual disability, or a history of epilepsy
* Participants with an identified suicide risk, self-harm tendencies, or violent behavior

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Psychososcial Functioning | 3 months
  Psychosocial functioning refers to an individual's ability to interact with their environment and to perform effectively in various social roles, such as being an employee, student, spouse, family member, or friend. This definition also encompasses individuals' capacity to fulfill these roles, engage in self-care, and derive satisfaction from leisure and recreational activities.
  In order to measure psychososcial functioning in detail, Social Functioning Scale (SFS) was used. SFS is a self-report scale that aims to measure social functioning in schizophrenia considering the period of last three months. The scale has seven specific areas of social functioning including social engagement/withdrawal, interpersonal behavior, recreation, pro-social activities, independence-performance, independence-competence and employment.
Psychosocial Functioning | 4 weeks
  In order to measure psychosocil functioning, Personal and Social Performance Scale (PSP) was used. PSP is an interview-based evaluation scale. It provides an assessment in functioning across four dimensions including socially useful activities, personal and social relationships, self-care, disturbing and aggressive behaviors. Each dimension is rated at six levels (absent, mild, manifest but not marked, marked, severe, very severe). Although each dimension is rated individually, a single score of social functioning is obtained ranging from 0 to 100. Higher score indicates better functioning.

SECONDARY OUTCOMES:
Sense of Presence | 1 week
  Sense of presence refers to 'being in the environment'. Virtual reality environments require a relative level of sense of presence to provide immersive effect. Sense of presence is measured in cVR-PTP group in a weekly basis after each session. Sense of presence was measured by using Presence Questionnaire (PQ). It is a Likert-type self-report scale with a five-factor structure: involvement, adaptation/immersion, sensory fidelity, interface quality and interaction. Participants who have experienced a virtual reality environment rate each item on a scale from 1 (not at all) to 5 (completely). The scale was originally developed by Witmer et al.

CONTACTS AND LOCATIONS:
Overall Officials: Köksal Alptekin, MD, Professor, Principal Investigator — Dokuz Eylul University; Faik Kartelli, PhD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Psychiatry, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this study will be shared upon reasonable request to the corresponding author, beginning after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Background] Bell, I.H., Pot-Kolder, R., Rizzo, A. et al. Advances in the use of virtual reality to treat mental health conditions. Nat Rev Psychol 3, 552-567 (2024). https://doi.org/10.1038/s44159-024-00334-9
- [Background] Witmer B. G., Jerome C. J. and Singer M. J. , "The Factor Structure of the Presence Questionnaire," in Presence, vol. 14, no. 3, pp. 298-312, June 2005, doi: 10.1162/105474605323384654.
- [Background] Priebe S. Social outcomes in schizophrenia. Br J Psychiatry Suppl. 2007 Aug;50:s15-20. doi: 10.1192/bjp.191.50.s15. PMID 18019039
- [Background] Bosc M. Assessment of social functioning in depression. Compr Psychiatry. 2000 Jan-Feb;41(1):63-9. doi: 10.1016/s0010-440x(00)90133-0. PMID 10646621
- [Background] Schroeder AH, Bogie BJM, Rahman TT, Therond A, Matheson H, Guimond S. Feasibility and Efficacy of Virtual Reality Interventions to Improve Psychosocial Functioning in Psychosis: Systematic Review. JMIR Ment Health. 2022 Feb 18;9(2):e28502. doi: 10.2196/28502. PMID 35179501
- [Background] Wiebe A, Kannen K, Selaskowski B, Mehren A, Thone AK, Pramme L, Blumenthal N, Li M, Asche L, Jonas S, Bey K, Schulze M, Steffens M, Pensel MC, Guth M, Rohlfsen F, Ekhlas M, Lugering H, Fileccia H, Pakos J, Lux S, Philipsen A, Braun N. Virtual reality in the diagnostic and therapy for mental disorders: A systematic review. Clin Psychol Rev. 2022 Dec;98:102213. doi: 10.1016/j.cpr.2022.102213. Epub 2022 Oct 30. PMID 36356351